CLINICAL TRIAL: NCT07005219
Title: Efficacy of Minimal vs. Conventional Apical Preparation With Passive Ultrasonic Irrigation in Reducing Intracanal Bacteria: A Clinical Study
Brief Title: Efficacy of Apical Preparation With Passive Ultrasonic Irrigation in Reducing Intracanal Bacteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Melike Yavuz, Director, Clinical Research, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10840098-772.02-6513
Record Dates: First submitted 2025-05-22; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Periapical Periodontitis; Root Canal Infection
Keywords: apical periodontitis; irrigation activation; apical enlargement; ddPCR; bacterial species
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apical Enlargement with One Curve Mini #25/0.4 (Minimal Invasive Shaping) (Experimental): Intervention:
  * Root canal shaping using One Curve Mini #25/0.4 rotary file.
  * Irrigation with 3% NaOCl.
  * Passive Ultrasonic Irrigation (PUI) using IRRI S 21/25 tip on VDW Ultra device.
  * 3 cycles of ultrasonic activation (each 20 seconds, 1 ml NaOCl per cycle).
  * Ultrasonic tip placed 2 mm short of working length, without contacting canal walls.
  Interventions: Procedure: Root canal shaping with One Curve Mini #25/0.4 and passive ultrasonic irrigation
- Apical Enlargement with One Curve Mini #35/0.4 (Conventional Shaping) (Experimental): Intervention:
  * Root canal shaping using One Curve Mini #35/0.4 rotary file.
  * Irrigation with 3% NaOCl.
  * Passive Ultrasonic Irrigation (PUI) using IRRI S 21/25 tip on VDW Ultra device.
  * 3 cycles of ultrasonic activation (each 20 seconds, 1 ml NaOCl per cycle).
  * Ultrasonic tip placed 2 mm short of working length, without contacting canal walls.
  Interventions: Procedure: Root canal shaping with One Curve Mini #35/0.4 and passive ultrasonic irrigation

INTERVENTIONS:
Procedure: Root canal shaping with One Curve Mini #25/0.4 and passive ultrasonic irrigation — Participants in this group underwent root canal shaping using a One Curve Mini #25/0.4 rotary file. After mechanical preparation, passive ultrasonic irrigation (PUI) was performed using a VDW Ultra device with an IRRI S 21/25 ultrasonic tip. Irrigation was activated with 3% sodium hypochlorite (NaOCl) in three 20-second cycles, using 1 ml per cycle. The ultrasonic tip was placed 2 mm short of the working length without contacting canal walls.
  Arms: Apical Enlargement with One Curve Mini #25/0.4 (Minimal Invasive Shaping)
Procedure: Root canal shaping with One Curve Mini #35/0.4 and passive ultrasonic irrigation — Participants in this group underwent root canal shaping using a One Curve Mini #35/0.4 rotary file. The same passive ultrasonic irrigation protocol was applied as in Arm 1, using 3% NaOCl in three 20-second cycles with 1 ml per cycle. The ultrasonic tip was positioned 2 mm short of the working length without contacting the canal walls.
  Arms: Apical Enlargement with One Curve Mini #35/0.4 (Conventional Shaping)

SUMMARY:
This study evaluates intracanal bacterial load in molar teeth with chronic apical periodontitis before and after root canal shaping with two different apical enlargement sizes and ultrasonic irrigation activation.

DETAILED DESCRIPTION:
This randomized controlled clinical trial investigated the effect of different apical enlargement sizes and passive ultrasonic irrigation (PUI) on the bacterial load in the mesial roots of mandibular molars diagnosed with chronic apical periodontitis. The study was conducted at Istanbul Medipol University Faculty of Dentistry, Endodontics Clinic, and included 24 patients who required primary root canal treatment and exhibited clinical and radiographic signs of chronic apical periodontitis.

Participants were randomly assigned to two groups (n=12 each). In Group 1, root canal shaping was performed using a One Curve Mini #25/0.4 rotary file. In Group 2, shaping was performed using a One Curve Mini #35/0.4 rotary file. In both groups, passive ultrasonic irrigation was applied using the VDW Ultra device with an IRRI S 21/25 ultrasonic tip. The irrigation protocol consisted of three 20-second cycles using 1 ml of 3% sodium hypochlorite (NaOCl) per cycle. The ultrasonic tip was positioned 2 mm short of the working length without contacting the canal walls.

Bacterial samples were collected from the mesial root canals during the treatment. The bacterial load was quantified using Droplet Digital PCR (ddPCR), a highly sensitive and precise molecular technique that allows absolute quantification of bacterial DNA. This method was chosen because it enables accurate detection of bacterial reduction following the interventions.

ELIGIBILITY:
Inclusion Criteria

* a non-contributory medical history
* must have an asymptomatic mandibular molar with periapical lesions of>2.0x2.0 mm around the mesial roots
* must be diagnosed as chronic apical periodontitis

Exclusion Criteria

* Patients with acute clinical symptoms
* Teeth with previous root canal treatment
* non-restorable teeth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-02-24 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Reduction in Bacterial Load | During operation.
  Quantitative reduction in bacterial load in the mesial root canals of mandibular molars with apical periodontitis, as measured by Droplet Digital PCR (ddPCR), following different apical enlargement sizes and passive ultrasonic irrigation activation, provides quantitative data that can be statistically analyzed to compare the two intervention groups (#25/0.4 vs. #35/0.4 apical enlargement).

CONTACTS AND LOCATIONS:
Overall Officials: Melike Yavuz, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Esenler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After its publication in a journal, we want to share our data.
Supporting Information: Study Protocol, SAP
Time Frame: After its publication in a journal, we want to share our data.

REFERENCES:
- [Derived] Yavuz M, Eyuboglu TF, Eroglu SE, Hepsenoglu YE. The effect of apical preparation size and passive ultrasonic activation on microbial load in root canals with periapical lesions. Sci Rep. 2025 Dec 6;16(1):1264. doi: 10.1038/s41598-025-30950-1. PMID 41350378